CLINICAL TRIAL: NCT06568458
Title: A Phase 1, 3-Part, Open-label Study to Assess the Pharmacokinetic Interaction Between BMS-986278 and Nintedanib, the Relative Bioavailability of BMS-986278 Tablet Formulations, and the Food Effect on the Pharmacokinetics of BMS-986278 When Orally Administered as a Phase 3 Tablet Formulation in Healthy Participants
Brief Title: A Study to Assess the Extent of Drug Interaction Between BMS-986278 and Nintedanib, the Relative Bioavailability of BMS-986278 in Tablet and the Effect That Food Has on BMS-986278 in Tablet Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM027-1026
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part I: Period A (Experimental)
  Interventions: Drug: Nintedanib
- Part I: Period B (Experimental)
  Interventions: Drug: BMS 986278
- Part I: Period C (Experimental)
  Interventions: Drug: Nintedanib; Drug: BMS 986278
- Part II: Period 1 (Experimental)
  Interventions: Drug: BMS 986278
- Part II: Period 2 (Experimental)
  Interventions: Drug: BMS 986278
- Part II: Period 3 (Experimental)
  Interventions: Drug: BMS 986278
- Part III: Period 1 (Experimental)
  Interventions: Drug: BMS 986278
- Part III: Period 2 (Experimental)
  Interventions: Drug: BMS 986278

INTERVENTIONS:
Drug: Nintedanib — Specified Dose on specified days
  Arms: Part I: Period A; Part I: Period C
Drug: BMS 986278 — Specified dose on specified days
  Arms: Part I: Period B; Part I: Period C; Part II: Period 1; Part II: Period 2; Part II: Period 3; Part III: Period 1; Part III: Period 2

SUMMARY:
The Purpose of the Study is to Assess the Drug Interaction and Bioavailability of BMS-986278 in Tablet Formulations and the Effect that Food has on BMS-986278 in Tablet Formulation in Healthy Participants

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy males and females (INOCBP)
* Participant must have Body mass index (BMI) of 18.0 kg/m2 through 32.0 kg/m2, inclusive.
* Participant must have Body weight ≥ 50 kg

Exclusion Criteria:

* Participant must not have current or recent GI disease
* Participant with evidence of organ dysfunction or any clinically significant deviation, as determined by investigator, from normal in physical examination, vital signs, 12-lead ECG, or clinical laboratory determinations beyond what is consistent with the target population.
* Participant with prior exposure to BMS-986278 and exposure of any investigational drug or placebo within 4 weeks of study intervention administration.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Days 4, 17, 21 (Part-1); Days 1, 7, 13 (Part-2); Days 1, 7 (Part-3)
Area under the plasma concentration-time curve within a dosing interval AUC(TAU) | Day 4, 17 and 21 of Part 1
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration AUC(0-T) | Day 1-6 (part-2 and Part-3), Day 7-12 (Part2 and 3), Day 13-18) (Part-2)
Area under the plasma concentration-time curve from time zero extrapolated to infinite time AUC(INF) | Day 1-6 (part-2 and Part-3), Day 7-12 (Part2 and 3), Day 13-18) (Part-2)

SECONDARY OUTCOMES:
Number of participants with non-serious AEs (Adverse events) | Up to 28 Days post discontinuation of dosing
Number of participants with Serious AEs | Up to 28 Days post discontinuation of dosing
Number of participants with AEs leading to discontinuation | Up to 28 Days post discontinuation of dosing
Number of participants with Physical examination abnormalities | Up to 28 Days post discontinuation of dosing
Number of participants with vital sign abnormalities | Up to 28 Days post discontinuation of dosing
Number of participants with 12-lead electrocardiogram (ECG) abnormalities | Up to 28 Days post discontinuation of dosing
Number of participants with clinical laboratory abnormalities | Up to 28 Days post discontinuation of dosing
Time of maximum observed plasma concentration (Tmax) | Day 4, 17, 21 (Part-1), Day 1 (part-2 and Part-3), Day 7 (Part2 and 3), Day 13) (Part-2)
Apparent terminal phase half-life (T-HALF) | Day 1-6 (part-2 and Part-3), Day 7-12 (Part2 and 3), Day 13-18) (Part-2)
Apparent total body clearance (CLT/F) | Day 1-6 (part-2 and Part-3), Day 7-12 (Part2 and 3), Day 13-18) (Part-2)
Apparent volume of distribution of terminal phase (Vz/F) | Day 1-6 (part-2 and Part-3), Day 7-12 (Part2 and 3), Day 13-18) (Part-2)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com